CLINICAL TRIAL: NCT01494623
Title: Treating Working Memory Deficits in Patients With Schizophrenia Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Working Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 098 / 2006
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: working memory; schizophrenia; cognition; rTMS
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): Active treatment will be delivered at an intensity that is 90% of the RMT. Stimulation will be delivered at either 20 Hz or 10 Hz, depending on the patients' tolerance to the stimulation, with 50 stimulation trains of 30 stimuli each (i.e., 1500 stimuli) and an intertrain interval of 30 sec. 25 trains will be applied to to the left or right hemisphere followed by the other hemisphere.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but with only the side-edge resting on the scalp. The coil will be angled 45 degrees away from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Magnetic pulses to specified brain regions.
  Other Names: MagPro X100 Series (Medtronic A/S, Copenhagen, Denmark)

SUMMARY:
Deficits in working memory (WM) performance are the most significant cognitive impairments in schizophrenia (SCZ). It has also been shown that WM performance is contingent on the cortex synchronization, a process that relies on brain inhibition. Repetitive Transcranial Magnetic Stimulation (rTMS) has been demonstrated as an effective treatment for patients with SCZ and has been shown to increase brain inhibition and improve cognitive performance. In this study the investigators intend to:

* evaluate rTMS as a treatment for WM deficits in SCZ
* evaluate rTMS as a method to increase WM performance in healthy individuals
* determine if improvements in WM performance are related to enhanced synchronization of brain networks
* determine whether genetic polymorphisms predict cortical function and treatment response
* evaluate the influence of rTMS treatment on brain structure.

DETAILED DESCRIPTION:
To directly investigate whether enhanced gamma synchrony mediates rTMS enhancement of WM in patients with SCZ, and in healthy individuals the investigators propose the following study. The relationship between the improvements in WM performance and increased gamma synchrony following rTMS over the DLPFC will be investigated. Moreover, using statistical models, the investigators will further examine whether increased gamma synchrony mediates WM improvement in these patients. Therefore, in this study the investigators hope to clarify the neurophysiological mechanisms through which rTMS exerts its therapeutic effects on WM performance and develop rTMS as a novel therapeutic tool to enhance the treatment options available for one of the core cognitive deficits in this disorder.

There is considerable evidence to support the fact that WM deficits in schizophrenia are heritable and have a strong genetic component. This evidence emerges from genetic association studies, and studies demonstrating that unaffected relatives of schizophrenia patients also suffer WM deficits. Therefore, treatment response to rTMS may be at least partly contingent on genetic variation within each individual. In particular, GABAergic genes that code for GABAergic proteins which largely determine cortical inhibition may play a key role in treatment response to rTMS over the DLPFC. However, several other gene systems that interact with the GABAergic system may also play a role, and would also merit investigation. Similarly brain structure may also determine treatment response. For instance, volume or thickness of the DLPFC and DLPFC related circuitry has been shown to play a role in WM performance, and therefore, may be a biomarker of treatment response.

Objective 1: To improve WM in patients with SCZ, and in healthy individuals using rTMS.

Hypothesis 1:20 Hz rTMS over the DLPFC will be superior to sham stimulation in improving WM performance in patients with SCZ, and healthy individuals.

Objective 2: To evaluate if high frequency rTMS results in enhanced gamma synchrony SCZ and healthy individuals.

Hypothesis 2: 20 Hz rTMS over the DLPRC will be superior to sham stimulation at increasing gamma synchrony in patients with SCZ, and healthy individuals.

Objective 3: To determine if the rTMS induced increase in gamma band synchrony mediates the therapeutic effects of rTMS on WM performance in patients with SCZ and healthy individuals.

Hypothesis 3: Increased gamma band synchrony will be shown to mediate the therapeutic effects of rTMS on WM performance in SCZ and healthy individuals.

Objective 4: To test whether key polymorphisms in the GABAergic system, and related gene systems determine γ oscillatory activity and WM improvement following rTMS.

Hypothesis 4: GABAergic gene and related gene polymorphisms will determine variation in γ oscillatory activity and WM performance following rTMS treatment.

Objective 5: To examine whether brain structure is a biomarker of treatment response to rTMS Hypothesis 5: Increase in cortical thickness at DLPFC and in microstructural integrity in cortico-cortical white matter tracts connecting to DLPFC will correlate with n-back task performance after rTMS treatment.

ELIGIBILITY:
Inclusion Criteria for Schizophrenia Subjects:

* Voluntary and competent to consent
* SCID-IV Diagnosis of Schizophrenia or Schizoaffective Disorder
* Between the ages of 18 and 85

Inclusion Criteria for Healthy Subjects:

* voluntary and competent to consent
* between the ages of 18-85
* considered a healthy individual free of psychopathology based on the Personality Assessment Inventory
* right-handed determined by the TMS screening and demographic form
* self-reported non-smoker
* do not have a self-reported concomitant major medical or neurologic illness
* if a woman of childbearing potential, must be on an effective means of birth control determined through completion of the TMS screening and demographic form.

Exclusion Criteria for both Healthy Controls and Schizophrenia Subjects:

* Have a DSM-IV history of substance abuse or dependence in the last 6 months
* Have a concomitant major and unstable medical or neurologic illness
* Have a history of seizures
* Have a first degree relative with a history of a seizure disorder
* Are pregnant
* Have any clinically significant EEG activity indicating an increased risk of seizure, as confirmed by a neurologist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the performance on the N-back working memory task. | 4 weeks
  Specifically, we will evaluate if rTMS results in changes to the number of correct answers, omissions and errors as well as reaction times.

SECONDARY OUTCOMES:
Increase in gamma band synchrony | 4 weeks
  To ascertain whether high frequency rTMS is superior to sham stimulation in increasing gamma band synchrony our analysis will examine stimulus-locked changes in spectral power, phase, and coherence between electrodes.
Brain Imaging Changes | 4 weeks
  For brain imaging we will test for group differences using: (1) cortical thickness (2) volumetric measures, (3)diffusion based measures. Statistical tests measuring these differences will be conducted at baseline and at the conclusion of the study. We will control for possible effects of neuroleptic medication on MRI measures by regressing mean dosage levels multiplied by number of years on medication, for each of five classes of medication (typical neuroleptics, atypical neuroleptics, antiparkinsonian anticholinergics, lithium, benzodiazepines)

CONTACTS AND LOCATIONS:
Overall Officials: Z. Jeff Daskalakis, MD, PhD, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Barr MS, Farzan F, Rajji TK, Voineskos AN, Blumberger DM, Arenovich T, Fitzgerald PB, Daskalakis ZJ. Can repetitive magnetic stimulation improve cognition in schizophrenia? Pilot data from a randomized controlled trial. Biol Psychiatry. 2013 Mar 15;73(6):510-7. doi: 10.1016/j.biopsych.2012.08.020. Epub 2012 Oct 3. PMID 23039931
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research